CLINICAL TRIAL: NCT00757627
Title: Patient-reported Outcomes With Etoricoxib in Real Life
Brief Title: Patient-Reported Effectiveness and Safety of Etoricoxib in Osteoarthritis (OA)(0663-113)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0663-113; MK0663-113; 2008_029
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Results first posted 2010-05-11 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Etoricoxib

ARMS (1):
- 1 (Experimental): Etoricoxib
  Interventions: Drug: etoricoxib

INTERVENTIONS:
Drug: etoricoxib — etoricoxib 60 mg QD for 4 weeks.
  Other Names: Arcoxia

SUMMARY:
The purpose of this study is to collect disease burden of OA and the effectiveness and patient satisfaction of treatment by Etoricoxib in the normal practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Must Be Over 20 Years Of Age, Regardless Of Sex
* Must Have A Diagnosis Of OA That Requiring Treatment
* Patients Must Have Taken an NSAID, Cox-2 Or Opioids On The Majority Of Days During The Last 4 Weeks Before Enrollment Who Are Intolerant (Due To Gastrointestinal Adverse Events) Or Inadequately Respond To Current Therapy (Vas >= 40 mm On A Pain Scale From 0-100 mm)
* Excluding Osteoarthritis, The Patient Is Judged To Be In Otherwise General Good Health Based On Medical History, Physical Examination, And Routine Laboratory Tests
* Must Agree To Participate Voluntarily In The Study
* Must Have The Capacity To Understand And Answer The Questionnaires Used In The Study
* Must Agree To Return For A Follow-Up Visit With The Treating Physician Four Weeks After The Initiation Of Treatment With Etoricoxib
* Patient Is Willing To Sign Informed Consent Form

Exclusion Criteria:

* Under 20 Years Of Age
* Severe Hepatic Insufficiency (Child-Pugh Score > 9)
* Advanced Renal Insufficiency (Creatinine Clearance < 30 Ml/Min)
* Any Contraindication Or Warning Or Precaution As Mentioned In The Approved Study Drug Package Insert
* Gi Ulcer With Active Bleeding Present At Study Enrollment
* Patient Has A Recent History Of Stroke, Myocardial Infarction Or Transient Ischemic Attack (Within The Previous 2 Years)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lin HY, Cheng TT, Wang JH, Lee CS, Chen MH, Lei V, Lac C, Gammaitoni AR, Smugar SS, Chen WJ. Etoricoxib improves pain, function and quality of life: results of a real-world effectiveness trial. Int J Rheum Dis. 2010 May;13(2):144-50. doi: 10.1111/j.1756-185X.2010.01468.x. PMID 20536599

RESULTS

PARTICIPANT FLOW:
Groups:
- Etoricoxib: Etoricoxib 60 mg once a day (q.d.)
Period: Overall Study
Arm/Group | Etoricoxib
Started | 500
Completed | 419
Not Completed | 81
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 10
Not completed — Lost to Follow-up | 28
Not completed — Withdrawal by Subject | 27
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etoricoxib
Number analyzed (Participants) | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 365
  Male | 135
Patient-SF36 (Short form 36) domain scores [Mean (Standard Deviation); unit: Units on a scale] — SF36 consists of weighted scores of the 8 domains (physical functioning; role limitation due to physical problem; bodily pain; general health; vitality; social functioning; role limitation due to emotional problem; mental health), each is measured with scale score ranged from 0≈100, with 100 representing the best possible functioning).
  Units on a scale
    SF-36 Physical functional | 45.1 (51.3)
    SF-36 Role limitation due to physical problem | 24.0 (42.5)
    SF-36 Bodily pain | 52.4 (63.9)
    SF-36 General health | 52.7 (54.5)
    SF-36 Vitality | 55.9 (57.6)
    SF-36 Social functioning | 69.0 (78.3)
    SF-36 Role limitation due to emotional problem | 41.3 (56.6)
    SF-36 Mental health | 61.7 (66.3)
TSQM (Treatment Satisfaction Questionnaire for Medication )domain scores [Mean (Standard Deviation); unit: Units on a scale] — TSQM consists of four domains (effectiveness; side effect; convenience and overall satisfaction), domain scores ranged from 0(0=worst) to 100(100=best) were derived from converting the original Likert's scales to VAS scale.
  Units on a scale
    TSQM - Effectiveness | 52.1 (55.6)
    TSQM - Side effect | 56.9 (55.7)
    TSQM - Convenience | 68.0 (68.8)
    TSQM - Overall satisfaction | 44.1 (45.7)
The mean of patient BPI (Brief Pain Inventory) scores [Mean (Standard Deviation); unit: Units on a scale] — BPI consists of pain and pain interference domains. For pain (0=no pain to 10=extreme pain); for Interference ( 0=no interference to 10= greatest interference).
  Units on a scale
    BPI -Worst pain | 6.4 (4.9)
    BPI -Least pain | 3.2 (2.5)
    BPI-Average pain | 4.9 (3.8)
    BPI -Pain right now | 4.4 (3.1)
    BPI -Interference on general activities | 2.9 (2.1)
    BPI - Mood | 3.2 (2.2)
    BPI -Walking | 4.3 (2.9)
    BPI - Normal work | 4.2 (2.9)
    BPI- Relations with other people | 2.5 (1.9)
    BPI - Sleep | 3.3 (2.3)
    BPI - Enjoyment of life | 3.0 (2.1)
The mean of patient WOMAC ( Western Ontario and McMaster Universities Osteoarthritis Index) subscale [Mean (Standard Deviation); unit: Units on a Scale] — The baseline domain scores of WOMAC included pain, stiffness, and difficult in doing daily activity. Each domain comprises of questions and VAS scales for scoring For pain domain, 0 represents no pain and 100 represents extreme pain; for stiffness domain, 0 represents no stiffness and 100 represents extreme stiffness; for difficult in doing daily activity domain, 0 represents no difficulty and 100 represents most difficulty.
  Units on a Scale
    WOMAC Pain subscale | 38.5 (22.9)
    WOMAC Stiffness subscale | 36.3 (26.9)
    WOMAC Physical Function subscale | 38.0 (24.8)

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline in Patient WOMAC Domain Scores at Week 4
Description: The change from baseline in 3 domain scores (pain, stiffness, and difficult in doing daily activity) of WOMAC at week 4 were measured. Each domain comprises of questions and VAS scales for scoring. For pain domain, 0 represents no pain and 100 represents extreme pain; for stiffness domain, 0 represents no stiffness and 100 represents extreme stiffness; for difficult in doing daily activity domain, 0 represents no difficulty and 100 represents most difficulty.
Time Frame: Baseline and Week 4
Population: Only patients with baseline and week 4 data were included in this analysis of change
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Etoricoxib: Etoricoxib 60 mg q.d.
Arm/Group | Etoricoxib
Number analyzed (Participants) | 418
Units on a Scale
  WOMAC Pain subscale (n=418) | -10.0 (20.5)
  WOMAC Stiffness subscale (n=418) | -7.9 (25.7)
  WOMAC Physical Function subscale (n=416) | -8.0 (19.6)

2. Secondary Outcome: Physicians' Global Assessment of Patients' Response to Therapy at Baseline Using IGART (Investigator Global Assessment of Response to Therapy)
Description: The IGART comprised of five categories: No response, poor response, fair response, good response, and excellent response. The percentage of participants who met the criteria of any of the 5 categories at baseline were collected.
Time Frame: Baseline
Population: Only patients with baseline and week 4 data were included.
Measure: Number; unit: Percentage of Participants
Groups:
- Etoricoxib (Baseline): Etoricoxib 60 mg q.d.
Arm/Group | Etoricoxib (Baseline)
Number analyzed (Participants) | 500
Percentage of Participants
  No Response | 4.40
  Poor Response | 57.60
  Fair Response | 36.40
  Good Response | 1.60
  Excellent Response | 0.00

3. Secondary Outcome: Physicians' Global Assessment of Patients' Response to Therapy at Week 4 Using IGART
Description: The IGART comprised of five categories: No response, poor response, fair response, good response, and excellent response. The percentage of participants met the criteria of any of the 5 categories at week 4 were collected.
Time Frame: Week 4
Population: Per Protocol
Measure: Number; unit: Percentage of Participants
Groups:
- Etoricoxib (Week 4): Etoricoxib 60 mg q.d.
Arm/Group | Etoricoxib (Week 4)
Number analyzed (Participants) | 430
Percentage of Participants
  No response | 5.81
  Poor response | 16.05
  Fair response | 35.35
  Good response | 36.74
  Excellent response | 6.05

4. Primary Outcome: The Percentage of Participants Achieving ≥30% Decrease From Baseline in Pain Intensity as Measured by WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) Question 1 "Pain Walking on a Flat Surface" at Week 4
Description: WOMAC for pain assessment by patient (0-100 mm Visual Analog Scale (VAS) with 0 represent "no pain" and 100 represent "extreme pain")
Time Frame: Baseline and end of week 4
Population: Per protocol (all patients who completed the WOMAC"pain walking on a flat surface " question at baseline and follow up visit at week 4 will be included for analysis of this endpoint.
  Among the 419 patients with follow up visit data, 27 patients rated 0 in their VAS pain score at baseline and were excluded from this analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etoricoxib
Number analyzed (Participants) | 392
Percentage of Participants | 52.04

5. Secondary Outcome: Patient Assessment of General Health Outcome by EuroQoL-5 Dimensions (EQ-5D) at Baseline
Description: The percentage of participants who met the criteria of any of the 3 categories of EQ-5D at baseline and at week 4 were collected.The EQ-5D comprises of 5 dimensions (mobility, self-care, usual activities, pain / discomfort, and anxiety / depression) to be answered using a 3-categorical Likert's scales of: [No problem, Some problem, and Not able to carry out] for mobility, self-care and usual activities and [Not present, moderate and extreme] for discomfort and anxiety/depression.
Time Frame: Baseline
Population: Only patients with baseline and week 4 data were included in the analysis.
  Week 4 N Values; Motility 423 , Self care 422 , Daily Activity 421 , Pain/Discomfort 421 , Anxiety/Depressed 422
Measure: Number; unit: Percentage of Participants
Arm/Group | Baseline - EQ-5D
Number analyzed (Participants) | 500
Percentage of Participants
  Motility (n=499) No problem | 54.91
  Motility (n=499) Some problem | 45.09
  Motility (n=499) Not able to carry out | 0.00
  Self care (n=499) No problem | 86.97
  Self care (n=499) Some problem | 12.63
  Self care (n=499) Not able to carry out | 0.40
  Daily activity (n=499) No problem | 54.91
  Daily activity (n=499) Some problem | 43.69
  Daily activity (n=499) Not able to carry out | 1.40
  Pain/Discomfort (n=500) Not present | 10.00
  Pain/Discomfort (n=500) Moderate | 79.60
  Pain/Discomfort (n=500) Extreme | 10.40
  Anxiety/Depressed (n=500) Not present | 51.60
  Anxiety/Depressed (n=500) Moderate | 44.00
  Anxiety/Depressed (n=500) Extreme | 4.40

6. Secondary Outcome: Patient Assessment of General Health Outcome by EuroQoL-5 Dimensions (EQ-5D) at Week 4
Description: The percentage of participants who met the criteria of any of the 3 categories of EQ-5D at baseline and at week 4 were collected.The EQ-5D comprises of 5 dimensions (mobility, self-care, usual activities, pain / discomfort, and anxiety / depression) to be answered using a 3-categorical Likert's scales of: [No problem, Some problem, and Not able to carry out] for mobility, self-care and usual activities and [ Not present, moderate and extreme]for discomfort and anxiety/depression
Time Frame: Week 4
Population: per protocol
Measure: Number; unit: Percentage of participants
Arm/Group | Week 4 - EQ-5D
Number analyzed (Participants) | 423
Percentage of participants
  Motility (n=423) No problem | 67.61
  Motility (n=423) Some problem | 32.39
  Motility (n=423) Not able to carry out | 0.00
  Self care (n=422) No problem | 90.05
  Self care (n=422) Some problem | 9.48
  Self care (n=422) Not able to carry out | 0.47
  Daily activity (n=421) No problem | 61.76
  Daily activity (n=421) Some problem | 37.29
  Daily activity (n=421) Not able to carry out | 0.95
  Pain/Discomfort (n=421) Not present | 23.04
  Pain/Discomfort (n=421) Moderate | 73.63
  Pain/Discomfort (n=421) Extreme | 3.33
  Anxiety/Depressed (n=422) Not present | 61.37
  Anxiety/Depressed (n=422) Moderate | 36.97
  Anxiety/Depressed (n=422) Extreme | 1.66

7. Secondary Outcome: Change From Baseline of Patient BPI (Brief Pain Inventory) Scores at Week 4
Description: BPI consists of pain and pain interference domains. For pain (0=no pain to 10=extreme pain); for pain interference ( 0=no interference to 10= greatest interference).
Time Frame: Baseline and Week 4
Population: Only patients with both baseline and week 4 follow up data were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Etoricoxib
Number analyzed (Participants) | 419
Units on a Scale
  BPI Worst pain (n=418) | -1.5 (2.4)
  BPI Least pain (n=417) | -0.6 (2.2)
  BPI Average pain (n=419) | -1.0 (2.0)
  BPI Pain right now (n=416) | -1.3 (2.6)
  BPI Interference on general activities (n=419) | -0.8 (2.5)
  BPI Interference on Mood (n=419) | -1.0 (2.7)
  BPI Interference on Walking (n=419) | -1.2 (2.5)
  BPI Interference on Normal work (n=419) | -1.1 (2.8)
  BPI Interference on Relations (n=418) | -0.6 (2.6)
  BPI Interference on Sleep (n=419) | -1.0 (2.8)
  BPI Interference on Enjoyment of life(n=419) | -0.8 (2.7)

8. Secondary Outcome: Changes From Baseline in Patient TSQM (Treatment Satisfaction Questionnaire for Medication) Domain Scores at Week 4
Description: TSQM consists of four domains (effectiveness; side effect; convenience and overall satisfaction), domain scores ranged from 0 (0=worst) to 100 (100=best) were derived from converting the original Likert's scales to VAS scale.
Time Frame: Baseline and Week 4
Population: 22 patients who reported side effects at baseline and week 4 were included in "side effect" evaluation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Etoricoxib
Number analyzed (Participants) | 419
Units on a Scale
  Effectiveness ((n=418) | 2.8 (17.0)
  Side Effect (n=22) | -3.8 (16.4)
  Convenience (n=418) | 0.9 (10.8)
  Overall (n=419) | 1.1 (20.9)

9. Secondary Outcome: Change From Baseline in Number of Days Patient Miss From Work or House Keeping Work at Week 4
Time Frame: Baseline and Week 4
Population: Only patients with both baseline and week 4 data were included in this analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Etoricoxib
Number analyzed (Participants) | 411
Days
  Days Missed From Work (n=138) | -0.4 (1.6)
  Days Missed From Housekeeping Work (n=411) | -2.3 (6.8)

10. Secondary Outcome: Change From Baseline in Patient-SF36 (Short Form 36) Domain Scores at Week 4
Description: Weighted scores of the 8 domains of SF36 (i.e., physical functioning; role limiting due to physical problem; bodily pain; general health; vitality; social functioning; role limiting due to emotional problem; mental health) were scored on a scale from 0 ~100, with 100 representing the best possible functioning)
Time Frame: Baseline and Week 4
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Etoricoxib 60 mg q.d.
Number analyzed (Participants) | 419
Units on a Scale
  SF36 Physical Functioning (n=418) | 5.2 (19.9)
  SF36 Role Limiting Due to Physical Problem (n=418) | 17.6 (49.3)
  SF36 Bodily Pain (n=418) | 10.6 (17.7)
  SF36 General Health (n=419) | 2.0 (16.2)
  SF36 Vitality (n=417) | 1.4 (15.1)
  SF36 Social Functioning (n=419) | 8.7 (20.3)
  SF36 Role Limiting Due to Emotional Problem(n=418) | 14.0 (50.4)
  SF36 Mental Health (n=417) | 4.4 (14.0)

ADVERSE EVENTS:
Time Frame: From baseline to end of week 4
Arm/Group | Etoricoxib
Serious Adverse Events (participants affected / at risk) | 6/500
Other Adverse Events (participants affected / at risk) | 82/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib (N=500)
Peritoneal adhesion (Gastrointestinal disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Lung abscess, chest pain/tightness and tremor (General disorders) | 1 (1)
Traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Urethritis (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib (N=500)
Abdominal distension / flatulence (Gastrointestinal disorders) | 6 (6)
Abdominal pain, upper (Gastrointestinal disorders) | 6 (6)
Dizziness (Nervous system disorders) | 11 (12)
Edema , face/eye /hand/leg (Vascular disorders) | 24 (24)
Headache (Nervous system disorders) | 5 (5)
Hypertension / elevated blood pressure (Vascular disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 6 (6)
Palpitation (Cardiac disorders) | 8 (8)
Skin rash (Skin and subcutaneous tissue disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
Open-labeled, non-controlled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.